CLINICAL TRIAL: NCT01581671
Title: Non-Invasive Peripheral Arterial Tonometry (EndoPAT) Increases Diagnostic Yield of Coronary Artery Disease by Coronary Angiography
Brief Title: Non-Invasive EndoPAT Increases Diagnostic Yield of CAD by Coronary Angiography
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Itamar-Medical, Israel (Industry)
Responsible Party: Principal Investigator, Amir Lerman, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 10-005160
Record Dates: First submitted 2011-11-22; First posted 2012-04-20 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients having a first time angiogram: Patients who are coming to the Cardiac Cath Lab to have an angiogram for the first time

SUMMARY:
The purpose of this study is to assess the non-invasive, Peripheral Arterial Tonometry (PAT) testing as another way of predicting potential coronary artery blockages in the heart.

DETAILED DESCRIPTION:
We are conducting a 16 minute, non-invasive EndoPAT test on patients coming to our cath lab for a first-time angiogram. The angiogram results will be compared to the EndoPAT results to determine if the EndoPAT test, which generates a score, is successful in predicting who may have blockages in their coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patients without known coronary disease who are referred for coronary angiography.
* Adults 18 years and older.

Exclusion Criteria:

* Patients with known coronary disease, acute coronary syndrome, cardiac transplantation, and severe connective tissue disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming to the Cardiac Cath Lab to determine if they have coronary artery disease
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine if the assessment of endothelial function by non-invasive peripheral arterial tonometry improves diagnostic yield of elective coronary angiography | same day as the angiogram
  Will compare the score of the EndoPAT test to the outcome of the angiogram to determine if the score is predictive of coronary artery disease.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, B.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States